CLINICAL TRIAL: NCT02571816
Title: A Phase 1 Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of ASP2215
Brief Title: A Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of ASP2215
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2215-CL-0106
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Hepatic Impairment; Healthy
Keywords: Hepatic Impairment; Mild Hepatic Impairment; Healthy; ASP2215; Moderate Hepatic Impairment
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP2215: Subjects with mild hepatic impairment (Experimental): Subjects with Child Pugh classification score of 5-6 (mild)
  Interventions: Drug: ASP2215
- ASP2215: Subjects with moderate hepatic impairment (Experimental): Subjects with Child Pugh classification score of 7-9 (moderate)
  Interventions: Drug: ASP2215
- ASP2215: Subjects with normal hepatic function (Experimental): Healthy subjects that match with respect to age, sex and body mass index (BMI)
  Interventions: Drug: ASP2215

INTERVENTIONS:
Drug: ASP2215 — oral

SUMMARY:
The purpose of this study is to compare the single-dose pharmacokinetics of ASP2215 in subjects with mild and moderate hepatic impairment to matched healthy subjects with normal hepatic function.

This study will also assess the safety and tolerability of single-dose ASP2215 in subjects with mild and moderate hepatic impairment and matched control subjects.

DETAILED DESCRIPTION:
Subjects will be admitted to the site one day before each study drug administration (i.e. Day -1) and confined at the site till the collection of post-dose PK samples (Day 21). For subjects with hepatic impairment, subject will discharge on Day 21, and will visit the clinical unit on Day 24 (±1 day) and Day 28 (±1 day) for collection of post-dose PK samples. End of study Visit For Healthy subjects will take place 1 to 5 days following collection of last PK sample.

ELIGIBILITY:
Inclusion Criteria:

A prospective subject is eligible for the clinical study if all of the following apply:

* Subject has a Body Mass Index (BMI) range of 18.5 - 34.0 kg/m2, inclusive and weighs at least 50 kg at screening.
* Female subject must be nonchildbearing potential;

  * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
  * Documented surgically sterile (at least 1 month prior to screening), and
  * Female subject must have a negative pregnancy test at screening and Day -1.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 45 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 45 days after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using 2 forms of highly effective birth control (1 of which must be a barrier method) starting at screening and continue throughout the study period and for 105 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 105 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the last study visit.

In addition, subjects with mild or moderate hepatic impairment must also meet the following inclusion criterion:

* Subject must have a Child-Pugh classification Class A (mild, 5 to 6 points) or Class B (moderate, 7 to 9 points) liver function impairment at screening.

Exclusion Criteria:

A prospective subject will be excluded from participation in this clinical study if any of the following apply:

* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP2215, or any components of the formulation used.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies prior to study drug administration).
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has a long QT interval (QTc) at baseline
* Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or long corrected QT interval (QTc) syndrome or family history of long QTc syndrome
* Subjects with hypokalemia and hypomagnesemia at screening (defined as values below lower limit of normal).
* Subject has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure (SBP) >160 mmHg; mean diastolic blood pressure (DBP) >100 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) at day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject who has received the following drugs/products within 2 weeks prior to dosing:

  * Strong or moderate inhibitors (e.g., ketoconazole or fluconazole) or inducers (e.g., rifampin or phenytoin) of cytochrome P450 (CYP)3A4
  * Inhibitors and inducers of P-glycoprotein (P-gp)
  * Substrates of multidrug and toxin extrusion (MATE) 1
  * Drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5 hydroxytryptamine receptor 2B (5HT2BR)
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse at screening or day -1 (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates).
* Subject has used any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject anticipates an inability to abstain from xanthine (e.g., caffeine), grapefruit, Seville oranges (including marmalade), star fruit or any products containing these items from 72 hours prior to day -1 and throughout the duration of the study.
* Subject has significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has participated in any clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for study participation.
* Subject is an employee of the Astellas Group or Contract Research Organization.

In addition, healthy subjects must also NOT meet the following exclusion criteria:

* Subject used any prescribed or nonprescribed drugs (including vitamins, oral contraceptives or hormone replacement therapy, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of acetaminophen (up to 2 g per day).
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol defined clinical laboratory tests at screening or day -1.
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, hepatitis B core antibody or human immunodeficiency virus type 1 or 2 at screening.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the investigator.
* Subject has any of the liver chemistry tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase and total bilirubin) above the upper limit of normal at day -1. If the test is outside the reference range, the test may be repeated once.

In addition, subjects with mild or moderate hepatic impairment must also NOT meet the following exclusion criteria:

* Subject has any clinically significant abnormality, not related to their current disease state, following the investigator's review of the physical examination, ECG and protocol defined clinical laboratory tests at screening or day -1.
* Subject has a fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period (e.g., worsening ascites, infection of ascites, fever, active gastrointestinal bleeding).
* Subject has had a change in dose regimen of medically required medication within the last 2 weeks before prestudy examination (allowed co medication in patients), and/or the use of unallowed co medication in the 3 weeks prior to admission to the clinical unit (not allowed: any known hepatic enzyme altering agents or compounds known to restrict metabolism).
* Subject has presence of a hepatocellular carcinoma or an acute liver disease caused by an infection or drug toxicity.
* Subject has severe portal hypertension or surgical porto-systemic shunts, including Transjugular intrahepatic portosystemic shunt (TIPSS).
* Subject has biliary liver cirrhosis, biliary obstruction or other cause of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Subject has signs of significant hepatic encephalopathy (hepatic encephalopathy grade >2).
* Subject has severe ascites and/or pleural effusion.
* Subject had esophageal/gastric variceal bleeding in the past 6 months prior to screening.
* Subject has a thrombocyte level below 40 × 109 /L and/or hemoglobin below 90 g/L.
* Subject had a previous liver transplantation.
* Subject has severe or moderate renal dysfunction (estimated glomerular filtration rate [eGFR] below 60 mL/min/1.73m2) estimated via the following Modification of Diet in Renal Disease (MDRD) equation: eGFR (mL/min/1.73 m2) = 175 × (SCr [mg/dL]) -1.154 × (Age) -0.203 × (0.742 if female) × (1.212 if black)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-03-05 (Actual); Study Completion 2016-03-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP2215 in plasma: AUCinf | Up to Day 28
  Area under the curve from time zero to infinity (AUCinf)
Pharmacokinetics of ASP2215 in plasma: AUClast, 480 | Up to Day 28
  Area under the concentration-time curve from the time of dosing to the last measurable concentration within 480 hours postdose (AUClast,480)
Pharmacokinetics of ASP2215 in plasma: Cmax | Up to Day 28
  Maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics of ASP2215 in plasma: t1/2 | Up to Day 28
  Apparent Terminal Elimination Half-life (t1/2)
Pharmacokinetics of ASP2215 in plasma: tmax | Up to Day 28
  The time after dosing when Cmax occurs (tmax)
Pharmacokinetics of ASP2215 in plasma: CL/F | Up to Day 28
  Apparent total systemic clearance after extravascular dosing (CL/F)
Pharmacokinetics of ASP2215 in plasma: Vz/F | Up to Day 28
  Apparent volume of distribution during the terminal elimination phase after single extravascular dosing (Vz/F)
Pharmacokinetics of ASP2215 in plasma: fu | Up to Day 28
  Fraction of parent or metabolite available systemically unbound (=free fraction) (fu)
Pharmacokinetics of ASP2215 in plasma: AUClast | Up to Day 28
  Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast)
Pharmacokinetics of ASP2215 in plasma: AUClast,u | Up to Day 28
  Area under the concentration-time curve from the time of dosing to the last measurable concentration for unbound concentration (AUClast,u)
Pharmacokinetics of ASP2215 in plasma: AUCinf,u | Up to Day 28
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity for unbound concentration (AUCinf,u)
Pharmacokinetics of ASP2215 in plasma: AUClast,480,u | Up to Day 28
  Area under the concentration-time curve from the time of dosing to the last measurable concentration within 480 postdose for unbound concentration (AUClast,480,u)
Pharmacokinetics of ASP2215 in plasma: Cmax,u | Up to Day 28
  Maximum concentration for unbound concentration (Cmax,u)
Pharmacokinetics of ASP2215 in plasma: CLu/F | Up to Day 28
  Apparent total systemic clearance of unbound ASP2215 after extravascular dosing (CLu//F)
Pharmacokinetics of ASP2215 in plasma: Vz,u/F | Up to Day 28
  Apparent volume of distribution during the terminal elimination phase of unbound ASP2215 after extravascular dosing (Vz,u/F)
Safety profile assessed by Adverse Events (AEs), Clinical laboratory evaluations, 12-Lead electrocardiogram (ECG) and Vital signs | Up to Day 34
  Clinical laboratory evaluations include hematology, biochemistry, and urinalysis. Vital signs include oral temperature, respiration rate, pulse, and supine blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site US10001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] James AJ, Smith CC, Litzow M, Perl AE, Altman JK, Shepard D, Kadokura T, Souda K, Patton M, Lu Z, Liu C, Moy S, Levis MJ, Bahceci E. Pharmacokinetic Profile of Gilteritinib: A Novel FLT-3 Tyrosine Kinase Inhibitor. Clin Pharmacokinet. 2020 Oct;59(10):1273-1290. doi: 10.1007/s40262-020-00888-w. PMID 32304015
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=396